CLINICAL TRIAL: NCT03576495
Title: The Provider Awareness and Cultural Dexterity Toolkit for Surgeons Trial
Acronym: PACTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Howard University (Other); Johns Hopkins University (Other); Brown University (Other); Eastern Virginia Medical School (Other); Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Adil Haider, Kessler Director, Center for Surgery and Public Health, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P001237; 1R01MD011685-01A1 (NIH)
Record Dates: First submitted 2018-06-13; First posted 2018-07-03 (Actual); Results first posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Resident Knowledge and Attitudes Regarding Cross-cultural Care; Interpersonal and Communication Skills in Patient-clinician Encounters; Patient-reported Satisfaction With Resident Physicians Involved in Their Care; Patients' Clinical Health Outcomes After Surgery
Keywords: Medical education; Patient-reported satisfaction; Patient-reported outcomes; Cultural dexterity; Cross cultural care; Resident physician education

STUDY DESIGN:
Intervention Model Description: Sites will be assigned to an early intervention/retention assessment group or a delayed intervention group (control) for examination of the effectiveness of the intervention as well as learner retention.
Masking Description: Resident program directors and research staff will not be blinded to the implementation of curriculum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Intervention Group (Experimental): The investigators will assess the residents' knowledge, attitudes, and skills prior to and after the PACTS curriculum administration at half the sites (Early Intervention Group). Evaluation results in the Early Intervention Group will be compared to the Delayed Intervention (Active Comparator) group at time Period 2.
  Interventions: Other: PACTS curriculum
- Delayed Intervention Group (Active Comparator): The investigators will conduct baseline testing prior to the standard residency curriculum. These results will be compared to the Early Intervention Group (Experimental Group) at time period 2.
  Interventions: Other: Standard Residency Curriculum

INTERVENTIONS:
Other: PACTS curriculum — The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
  Arms: Early Intervention Group
Other: Standard Residency Curriculum — The standard residency curriculum consists of previously scheduled resident didactic sessions at all academic medical centers that may or may not include topics on cultural competency or cross-cultural care.
  Arms: Delayed Intervention Group

SUMMARY:
This study is designed to test the impact of a new curriculum, called Provider Awareness Cultural Dexterity Toolkit for Surgeons (PACTS), on surgical residents' cross-cultural knowledge, attitudes, and skills surrounding the care of patients from diverse cultural backgrounds, as well as clinical and patient-reported health outcomes for patients treated by surgical residents undergoing this training.

DETAILED DESCRIPTION:
In order to improve overall health outcomes of minority patients undergoing surgical care, the National Institute on Minority Health and Health Disparities (NIMHD) collaborated with the American College of Surgeons (ACS) and prioritized the evaluation and the the effect of improvement in culturally dexterous care on surgical outcomes for patients from disparity populations.

Poor outcomes in patients are attributed to poor patient-provider communication which may lead to treatment errors, inadequate pain management, less patient-centered care, decreased adherence to treatment plans, and worse overall clinical outcomes. Additionally, studies have shown that some surgeons have pro-White implicit biases, which are unconscious, automated preferences that individuals may not even be aware of.

Historically, formal training in cultural competency is generally integrated into medical education at the undergraduate level but it rarely continues up to the post-graduate level. Few surgical programs have attempted to incorporate cross-cultural communication skills into their educational paradigms, and the approaches to doing so have been inconsistent.

In order to add the surgical context in post-graduate level medical education, the investigators adopted a novel approach to cross-cultural communication for surgical trainees, known as cultural dexterity. Cultural dexterity refers to a set of skills and cognitive practices used to maximize communication across multiple dimensions of cultural diversity and deviates from the concept of cultural competency in that it does not demand that learners associate certain practices and behaviors with individuals based on generalizations.

Study design:

Cross-over, cluster-randomized trial

Study Procedures:

Curriculum Administration

The PACTS curriculum incorporates contemporary learning practices such as the "flipped classroom" model and team-based learning. It consists of e-learning modules and interactive sessions in which residents will apply concepts from the e-learning modules to role-play scenarios constructed in a team-based learning format. Residents will be given detailed, scripted prompts for the role-play sessions followed by structured feedback from peers and facilitators.

Outcome Measurement:

Residents

To evaluate the impact of PACTS on surgical residents' knowledge and attitudes about caring for diverse patients, the investigators will use a pre- and post-test in the form of validated instruments that assess knowledge, attitudes, and self-reported skills on a Likert-type scale.

Resident skills will also be objectively assessed through an Objective Structured Clinical Examination (OSCE) that will be created by the study staff and administered immediately before the intervention and 3 months after the intervention has been completed. The OSCE uses 5-point Likert scale questions to evaluate resident performance across multiple domains. These may be administered virtually or in-person.

A Standardized Patient evaluator and a third-party trained impartial observer will evaluate the residents on these domains, and the resulting numerical scores will be averaged. It will serve both a summative and educational purpose in this context.

Residents will be required to take a knowledge survey before and after receiving the PACTS curriculum or standard training. Attitudes regarding the importance of facing cross-cultural health care situations will be assessed across multiple domains using a novel survey instrument that is based on a survey that was used in a similar curriculum aimed at medical students, as well as the Values and Belief Systems domain.

Patients

To evaluate patients' satisfaction and clinical quality related to PACTS training, the investigators will administer surveys to patients treated by residents to determine satisfaction with pain management, communication, trust-building, and comprehension of the informed consent discussion two months before and after the intervention is implemented.

Patient satisfaction will be assessed using elements of the validated Patient Satisfactions Survey.

We plan to collect clinical surgical outcomes obtained from the National Surgical Quality Improvement Program (NSQIP) database for each patient participant before and after the PACTS curriculum is implemented to measure individual outcomes such as length of stay, postoperative complications, unplanned reoperations, and 30-day morbidity/mortality. A post hoc analysis of clinical outcomes will be performed.

ELIGIBILITY:
*Eligibility Criteria for Residents:

Inclusion Criteria:

- All residents in the general surgery program at Johns Hopkins University, Brigham and Women's Hospital, Brown University, Eastern Virginia Medical School, Massachusetts General Hospital, Beth Israel Deaconess Medical Center, Howard University, and Washington University in St. Louis.

Exclusion Criteria:

- Non-surgical residents at Johns Hopkins University, Brigham and Women's Hospital, Brown University, Eastern Virginia Medical School, Massachusetts General Hospital, Beth Israel Deaconess Medical Center, Howard University, and Washington University in St. Louis.

*Eligibility Criteria for Patients:

Inclusion Criteria:

* Admitted to surgical service under the care of a participating resident;
* Able to recognize resident as the main care provider from a photo;
* Able to consent as determined by a cognitive screen for capacity to give informed consent
* Fluent in English or Spanish.

Exclusion Criteria:

* Admitted to Intensive Care;
* Mentally impaired and/or not oriented to person/time/ place.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2901 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adil Haider, MD, MPH, Principal Investigator — Brigham and Women's Hospital; Douglas Smink, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (8):
- United States (8):
  - Howard University Hospital, Washington D.C., District of Columbia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - Rhode Island Hospital, Providence, Rhode Island
  - Eastern Virginia Medical School, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haider AH, Weygandt PL, Bentley JM, Monn MF, Rehman KA, Zarzaur BL, Crandall ML, Cornwell EE, Cooper LA. Disparities in trauma care and outcomes in the United States: a systematic review and meta-analysis. J Trauma Acute Care Surg. 2013 May;74(5):1195-205. doi: 10.1097/TA.0b013e31828c331d. PMID 23609267
- [Background] Haider AH, Scott VK, Rehman KA, Velopulos C, Bentley JM, Cornwell EE 3rd, Al-Refaie W. Racial disparities in surgical care and outcomes in the United States: a comprehensive review of patient, provider, and systemic factors. J Am Coll Surg. 2013 Mar;216(3):482-92.e12. doi: 10.1016/j.jamcollsurg.2012.11.014. Epub 2013 Jan 11. PMID 23318117
- [Background] Torain MJ, Maragh-Bass AC, Dankwa-Mullen I, Hisam B, Kodadek LM, Lilley EJ, Najjar P, Changoor NR, Rose JA Jr, Zogg CK, Maddox YT, Britt LD, Haider AH. Surgical Disparities: A Comprehensive Review and New Conceptual Framework. J Am Coll Surg. 2016 Aug;223(2):408-18. doi: 10.1016/j.jamcollsurg.2016.04.047. Epub 2016 Jun 10. No abstract available. PMID 27296524
- [Background] Cooper LA, Roter DL, Carson KA, Beach MC, Sabin JA, Greenwald AG, Inui TS. The associations of clinicians' implicit attitudes about race with medical visit communication and patient ratings of interpersonal care. Am J Public Health. 2012 May;102(5):979-87. doi: 10.2105/AJPH.2011.300558. Epub 2012 Mar 15. PMID 22420787
- [Background] Betancourt JR, Green AR, Carrillo JE, Ananeh-Firempong O 2nd. Defining cultural competence: a practical framework for addressing racial/ethnic disparities in health and health care. Public Health Rep. 2003 Jul-Aug;118(4):293-302. doi: 10.1093/phr/118.4.293. PMID 12815076
- [Background] Betancourt JR, Green AR, Carrillo JE, Park ER. Cultural competence and health care disparities: key perspectives and trends. Health Aff (Millwood). 2005 Mar-Apr;24(2):499-505. doi: 10.1377/hlthaff.24.2.499. PMID 15757936
- [Background] Horvat L, Horey D, Romios P, Kis-Rigo J. Cultural competence education for health professionals. Cochrane Database Syst Rev. 2014 May 5;2014(5):CD009405. doi: 10.1002/14651858.CD009405.pub2. PMID 24793445
- [Background] Weissman JS, Betancourt J, Campbell EG, Park ER, Kim M, Clarridge B, Blumenthal D, Lee KC, Maina AW. Resident physicians' preparedness to provide cross-cultural care. JAMA. 2005 Sep 7;294(9):1058-67. doi: 10.1001/jama.294.9.1058. PMID 16145026
- [Background] Shah SS, Sapigao FB 3rd, Chun MBJ. An Overview of Cultural Competency Curricula in ACGME-accredited General Surgery Residency Programs. J Surg Educ. 2017 Jan-Feb;74(1):16-22. doi: 10.1016/j.jsurg.2016.06.017. Epub 2016 Sep 20. PMID 27663082
- [Background] Haider AH, Dankwa-Mullan I, Maragh-Bass AC, Torain M, Zogg CK, Lilley EJ, Kodadek LM, Changoor NR, Najjar P, Rose JA Jr, Ford HR, Salim A, Stain SC, Shafi S, Sutton B, Hoyt D, Maddox YT, Britt LD. Setting a National Agenda for Surgical Disparities Research: Recommendations From the National Institutes of Health and American College of Surgeons Summit. JAMA Surg. 2016 Jun 1;151(6):554-63. doi: 10.1001/jamasurg.2016.0014. PMID 26982380
- [Derived] Allar BG, Ortega G, Chun MBJ, Rodriguez JGZ, Mullen JT, Lynch KA Jr, Harrington DT, Green AR, Lipsett PA, Britt LD, Haider AH, Smink DS, Kent TS; PACTS Trial Group. Changing Surgical Culture Through Surgical Education: Introduction to the PACTS Trial. J Surg Educ. 2024 Mar;81(3):330-334. doi: 10.1016/j.jsurg.2023.11.018. Epub 2023 Dec 23. PMID 38142149
- [Derived] Khubchandani JA, Atkinson RB, Ortega G, Reidy E, Mullen JT, Smink DS; PACTS Trial Group. Perceived Discrimination Among Surgical Residents at Academic Medical Centers. J Surg Res. 2022 Apr;272:79-87. doi: 10.1016/j.jss.2021.10.029. Epub 2021 Dec 20. PMID 34942508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of general surgery residents and surgical patients at Johns Hopkins University, Brigham and Women's Hospital, Brown University, and Eastern Virginia Medical School, Massachusetts General Hospital, Beth Israel Deaconess Medical Center, Howard University, and Washington University in St. Louis. We randomized at the site level to two groups: Early Intervention and Delayed Intervention. We reported our aggregate results for the residents and surgical patients in each group.
Pre-assignment Details: Inclusion criteria (Residents): All general surgery residents at all participating sites Exclusion criteria (Residents): All non-surgical residents at all participating sites
  Inclusion criteria (Patients): Admitted to a surgical service under the care of a participating resident with the capacity to give informed consent Exclusion criteria (Patients): Mentally impaired, admitted to intensive care
Units Other Than Participants: Residency Sites
Groups:
- Early Intervention Group: Residency sites (and in turn its residents) designated to the Early Intervention group will undergo assessment to evaluate residents' knowledge, attitudes, and skills prior to and after the PACTS curriculum administration. Follow-up testing will be conducted after one year to evaluate learner retention.
  Patients in the Early Intervention Group are patients who are cared for by a resident physician enrolled into the early intervention group, and monitors their patient satisfaction as well as clinical outcomes before and after the PACTS curriculum.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group: Residency sites and its participating residents designated to the delayed intervention group underwent baseline testing prior to the standard residency curriculum, and then received the PACTS curriculum the following year.
  Both between- and within-group differences will be examined based on curriculum exposure in intervention year 1 as well as within-group differences for the Delayed Intervention Group at the end of year 2.
  Patients designated to the Delayed Intervention Group are cared for by a resident physician enrolled into the delayed intervention group, and monitors their patient satisfaction as well as clinical outcomes before and after the PACTS curriculum.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
Period: Period 1 (0 Months)
Arm/Group | Early Intervention Group | Delayed Intervention Group
Started | 1489; 4 Residency Sites | 1412; 4 Residency Sites
Residents | 192; 4 Residency Sites | 214; 4 Residency Sites
Patients | 1297; 4 Residency Sites | 1198; 4 Residency Sites
Completed | 1438; 4 Residency Sites | 1372; 4 Residency Sites
Not Completed | 51; 0 Residency Sites | 40; 0 Residency Sites
Not completed — Lost to Follow-up | 51 | 40
Period: Period 2 (18 Months)
Arm/Group | Early Intervention Group | Delayed Intervention Group
Started | 1438; 4 Residency Sites | 1372; 4 Residency Sites
Residents | 141; 4 Residency Sites | 174; 4 Residency Sites
Patients | 1297; 4 Residency Sites | 1198; 4 Residency Sites
Completed | 1438; 4 Residency Sites | 1372; 4 Residency Sites
Not Completed | 0; 0 Residency Sites | 0; 0 Residency Sites
Period: Period 3 (36 Months)
Arm/Group | Early Intervention Group | Delayed Intervention Group
Started | 1438; 4 Residency Sites | 1372; 4 Residency Sites
Residents | 141; 4 Residency Sites | 174; 4 Residency Sites
Patients | 1297; 4 Residency Sites | 1198; 4 Residency Sites
Completed | 1438; 4 Residency Sites | 1372; 4 Residency Sites
Not Completed | 0; 0 Residency Sites | 0; 0 Residency Sites

BASELINE CHARACTERISTICS:
Population: A total of 8 residency sites were enrolled: 4 were designated to the Early Intervention group, and 4 were designated to the Delayed Intervention group. The baseline participants includes residents and patients.
Units Other Than Participants: Residency Sites
Groups:
- Early Intervention Group: Residency sites and its residents designated to the Early Intervention group will undergo assessment to evaluate residents' knowledge, attitudes, and skills prior to and after the PACTS curriculum administration. Follow-up testing will be conducted after one year to evaluate learner retention.
  Patients in the Early Intervention Group are patients who are cared for by a resident physician enrolled into the early intervention group, and monitors their patient satisfaction as well as clinical outcomes before and after the PACTS curriculum.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Total: Total of all reporting groups
Arm/Group | Early Intervention Group | Delayed Intervention Group | Total
Number analyzed (Participants) | 1438 | 1372 | 2810
Number analyzed (Residency Sites) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number of participants analyzed differs from the number enrolled due to loss to follow up.
  years
    Residents: number analyzed (Participants) | 141 | 174 | 315
    Residents | 30.1 (3.8) | 30.1 (3.8) | 30.1 (3.79)
    Patients: number analyzed (Participants) | 1297 | 1198 | 2495
    Patients | 55.24 (17) | 56.07 (17.3) | 55.64 (17.17)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The number of participants enrolled differed from the number analyzed due to loss to follow up.
  Participants
    Resident Sex/Gender: number analyzed (Participants) | 141 | 174 | 315
    Resident Sex/Gender: Male | 72 | 86 | 158
    Resident Sex/Gender: Female | 69 | 66 | 135
    Resident Sex/Gender: Non-Binary, Self-Describe, Not disclosed | 0 | 22 | 22
    Patient Sex/Gender: number analyzed (Participants) | 1297 | 1198 | 2495
    Patient Sex/Gender: Male | 670 | 605 | 1275
    Patient Sex/Gender: Female | 601 | 588 | 1189
    Patient Sex/Gender: Non-Binary, Self-Describe, Not disclosed | 26 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The number of participants analyzed differs from the number enrolled due to loss to follow up
  Participants
    Residents: number analyzed (Participants) | 141 | 174 | 315
    Residents: Hispanic or Latino | 15 | 10 | 25
    Residents: Not Hispanic or Latino | 123 | 119 | 242
    Residents: Unknown or Not Reported | 3 | 45 | 48
    Patients: number analyzed (Participants) | 1297 | 1198 | 2495
    Patients: Hispanic or Latino | 146 | 53 | 199
    Patients: Not Hispanic or Latino | 944 | 1020 | 1964
    Patients: Unknown or Not Reported | 207 | 125 | 332
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The number of participants analyzed differs from the number enrolled due to loss to follow up.
  Participants
    Residents: number analyzed (Participants) | 141 | 174 | 315
    Residents: White | 73 | 90 | 163
    Residents: Black | 23 | 11 | 34
    Residents: Asian | 28 | 20 | 48
    Residents: Multiracial/other | 17 | 14 | 31
    Residents: Not disclosed | 0 | 39 | 39
    Patients: number analyzed (Participants) | 1297 | 1198 | 2495
    Patients: White | 797 | 779 | 1576
    Patients: Black | 269 | 320 | 589
    Patients: Asian | 32 | 30 | 62
    Patients: Multiracial/other | 172 | 61 | 233
    Patients: Not disclosed | 27 | 8 | 35
Education [Count of Participants; unit: Participants] — Population: The number of analyzed differs from the number enrolled due to loss to follow up. The participants in the Early and Delayed Resident Groups are all physicians and therefore, are categorized as Master, Professional, and Doctorate degree level for education.
  Participants
    Residents: number analyzed (Participants) | 141 | 174 | 315
    Residents: No schooling, or completed to 1 or more years | 0 | 0 | 0
    Residents: Associates & Bachelors | 0 | 0 | 0
    Residents: Master, Professional, and Doctorate | 141 | 174 | 315
    Residents: Not disclosed | 0 | 0 | 0
    Patients: number analyzed (Participants) | 1297 | 1198 | 2495
    Patients: No schooling, or completed to 1 or more years | 700 | 634 | 1334
    Patients: Associates & Bachelors | 350 | 304 | 654
    Patients: Master, Professional, and Doctorate | 206 | 148 | 354
    Patients: Not disclosed | 41 | 112 | 153

OUTCOME MEASURES:

1. Primary Outcome: Change in Residents' Questionnaire Scores Measuring Knowledge From Pre- to Post-PACTS Curriculum
Description: The effect of PACTS curriculum on surgical residents' questionnaire scores measuring knowledge about caring for culturally diverse patients at time Period 2 (18 months). At this time, the Early Intervention Group had already received the PACTS curriculum. The Delayed Intervention Group had not received the PACTS curriculum, serving as the control group at this time period.
  Resident knowledge: Percent score out of 100, with range 0-100%. Higher values represent a better outcome, with 100% as the highest score possible. This is the average score for the Early Intervention and Delayed Intervention groups at Period 2.
Time Frame: Period 2 (18 months)
Population: Mean resident knowledge scores (from 0-100%) for surgical residents in both the Early Intervention and Delayed Intervention groups at Period 2 (18 months). Of the residents who completed the trial (141 for Early Intervention Group; 174 for Delayed Intervention Group), only 52 residents in the Early Intervention and 55 residents in the Delayed Intervention Group participated in the resident assessment at Period 2.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Early Intervention Group: The investigators will assess the residents' knowledge after the PACTS curriculum administration at half the sites (Early Intervention Group). Post-exposure effect in the Early Intervention Group was assessed at Period 2 (18 months).
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group: At 18 months (Period 2), resident knowledge was assessed using the standard residency curriculum.
Arm/Group | Early Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 52 | 55
score on a scale | 74.3 (8.96) | 71.7 (13.39)
Statistical Analysis 1: Comparison: Early Intervention Group vs Delayed Intervention Group; Test type: Superiority — We conducted a superiority statistical test to assess if residents' knowledge improved after exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum on resident knowledge, resident knowledge was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups; p = 0.2422, t-test, 2 sided — This p-value compares the average scores (in percent) of the residents' knowledge assessment at time period 2 between the Early Intervention and Delayed Intervention groups; Mean Difference (Final Values) = 2.6

2. Primary Outcome: Change in Residents' Cross Cultural Care Survey Scores From Pre- to Post-PACTS Curriculum
Description: The effect of PACTS curriculum on surgical residents' cross cultural care survey about caring for culturally diverse patients at time Period 2 (18 months). At this time period, the Early Intervention group received the PACTS curriculum, while the Delayed Intervention Group had not received the PACTS curriculum, serving as the control group. The cross cultural care survey was evaluated using a modified Likert type scale (with scale ranging from lowest to highest: very unprepared, somewhat unprepared, somewhat prepared, very well prepared). Resident scores were dichotomized into two groups, those reporting "very unprepared" and "somewhat unprepared", and those reporting "somewhat prepared" and "very well prepared." Here reported values are representative of the percentage of participants who reported "somewhat prepared" and "very well prepared" at time Period 2.
Time Frame: Period 2 (18 months)
Population: Percentage of residents who reported "somewhat prepared" and "very well prepared" for the cross cultural survey in both the Early Intervention and Delayed Intervention groups at time period 2. Of the residents who completed the trial (141 for Early Intervention Group; 174 for Delayed Intervention Group), only 52 residents in the Early Intervention and 55 residents in the Delayed Intervention Group completed the Cross Cultural Care Survey at Period 2.
Measure: Number; unit: percentage of participants
Groups:
- Early Intervention: The investigators will assess the residents' cross cultural care after administration of the PACTS curriculum (Early Intervention/Retention Group). Testing will be conducted after 18 months.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group: At 18 months (Period 2), resident cross cultural care was assessed after the standard residency curriculum.
Arm/Group | Early Intervention | Delayed Intervention Group
Number analyzed (Participants) | 52 | 55
percentage of participants | 88.2 | 88.2
Statistical Analysis 1: Comparison: Early Intervention vs Delayed Intervention Group; We conducted a superiority statistical test to assess if residents' preparation for caring for culturally diverse patients improved after exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum on resident preparedness assessed by the Cross-Cultural Care Survey, resident preparedness was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups; Test type: Superiority; p = 1.000, Chi-squared; Difference between percentage = 0

3. Primary Outcome: Change in Residents' Questionnaire Scores Regarding Self-Assessed Skills From Pre- to Post-PACTS Curriculum
Description: The effect of PACTS curriculum on surgical residents' self-assessed skills for caring for culturally diverse patients at time Period 2 (18 months). Self-assessed skills ranged from levels 1 to levels 4, with level 1 indicated less skilled, and level 4 indicating skillful. For purposes of comparison, resident scores were dichotomized into two groups: less skilled (referring to skill levels 1 and 2), and skillful (levels 3 and 4). Here reported values are representative of the percentage of participants who reported skill levels 3 or 4, indicating skillful. Results here demonstrate the proportion of residents in the Early Intervention (Intervention) group and Delayed Intervention (control group) who self-evaluated their skills as skillful at Period 2.
Time Frame: Period 2 (18 months)
Population: Of the residents who completed the trial (141 for Early Intervention Group; 174 for Delayed Intervention Group), only 52 residents in the Early Intervention and 55 residents in the Delayed Intervention Group participated in the questionnaire regarding self-assessed skills.
Measure: Number; unit: percentage of "skillful" participants
Groups:
- Early Intervention Group: The investigators will assess the residents' skills after the PACTS curriculum administration at Period 2 (18 months).
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group: At 18 months (Period 2), residents self-assessed skills were assessed after the standard residency curriculum.
Arm/Group | Early Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 52 | 55
percentage of "skillful" participants | 85.0 | 84.1
Statistical Analysis 1: Comparison: Early Intervention Group vs Delayed Intervention Group; We conducted a superiority statistical test to assess if residents' self-assessed skills improved after exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum on resident skills, resident skills were compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups; Test type: Superiority; p = 0.6295, Chi-squared; Percent difference = 0.9

4. Primary Outcome: Change in Residents' Questionnaire Scores Regarding Their Beliefs From Pre- to Post-PACTS Curriculum
Description: The effect of PACTS curriculum on surgical residents' beliefs regarding caring for culturally diverse patients at time Period 2 (18 months). At this time, the Early Intervention Group had already received the PACTS curriculum. The Delayed Intervention Group had not received the PACTS curriculum, serving as the control group at this time period. The questionnaire was scored using a modified Likert type scale with a range from lowest to highest: strongly disagree, moderately disagree, mildly disagree, strongly agree, moderately agree, mildly agree. Answers were dichotomized into two groups: strongly disagree, moderately disagree, and mildly disagree; and strongly agree, moderately agree, and mildly agree. Here reported values are representative of the proportion of participants who answered "strongly agree, moderately agree, and mildly agree."
Time Frame: Period 2 (18 months)
Population: Of the residents who completed the trial (141 for Early Intervention Group; 174 for Delayed Intervention Group), only 52 residents in the Early Intervention and 55 residents in the Delayed Intervention Group completed the questionnaire on beliefs at time Period 2.
Measure: Number; unit: percentage of participants
Groups:
- Early Intervention / Retention Group: The investigators will assess the residents' beliefs after the PACTS curriculum administration at half the sites (Early Intervention/Retention Group) at Time Period 2 (18 months).
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group: The investigators will evaluate surgical residents' beliefs regarding providing cross cultural care after the standard residency curriculum at 18 months (Period 2).
Arm/Group | Early Intervention / Retention Group | Delayed Intervention Group
Number analyzed (Participants) | 52 | 55
percentage of participants | 92.4 | 89.9
Statistical Analysis 1: Comparison: Early Intervention / Retention Group vs Delayed Intervention Group; We conducted a superiority statistical test to assess if residents' beliefs improved after exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum on resident beliefs, beliefs were compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups; Test type: Superiority; p = 0.0199, Fisher Exact; Difference between percentage = 2.5

5. Primary Outcome: Objective Structured Clinical Examination Scores
Description: Standardized Patient observers evaluated surgical residents on multiple dimensions of cultural dexterity and communication skills using Likert-type scales. The scale range, from lowest to highest was: "Not at all; a little bit; somewhat; mostly; a great deal." Scores were put into two groups: 1) not at all, a little bit, and somewhat; 2) mostly and a great deal. The percentage of residents who received scores of "mostly" and "a great deal" in categories of trust, limited english proficiency, consent, and pain were reported.
Time Frame: Period 2 (18 months)
Population: Of the residents who completed the trial (141 for Early Intervention Group; 174 for Delayed Intervention Group), only 59 residents in the Early Intervention and 111 residents in the Delayed Intervention Group completed the the OSCE at Period 2. Only 105 residents performed the OSCE on Limited English Proficiency in the Delayed Group
Measure: Number; unit: difference in the percentage
Groups:
- Early Intervention Group (Residents): Residents assigned to the Early Intervention group participated in Objective Structure Clinical Examinations where they are assessed by a Standardized Patient on dimensions of cultural dexterity and communication skills using Likert-type scales. Results from Period 2 (18 months) were after residents received the PACTS curriculum.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group (Residents): Residents assigned to the Delayed Intervention group participated in Objective Structure Clinical Examinations where they are assessed by a Standardized Patient on dimensions of cultural dexterity and communication skills using Likert-type scales. Results from Period 2 (18 months) were after residents received the standard curriculum.
Arm/Group | Early Intervention Group (Residents) | Delayed Intervention Group (Residents)
Number analyzed (Participants) | 59 | 111
difference in the percentage
  Limited English Proficiency/Informed Consent Period 2: number analyzed (Participants) | 59 | 105
  Limited English Proficiency/Informed Consent Period 2 | 60.9 | 63.1
  Trust/Pain Period 2 | 58.6 | 64.8
Statistical Analysis 1: Comparison: Early Intervention Group (Residents) vs Delayed Intervention Group (Residents); We conducted a superiority statistical test to assess if residents' OSCE performance improved after exposure to the PACTS curriculum. OSCE performance was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups. We compared the difference in the percentage of residents designated "mostly" and "a great deal" on Limited English Proficiency and Informed Consent OSCE; Test type: Superiority; p = 0.2665, Chi-squared; difference in the percentage = 2.2
Statistical Analysis 2: Comparison: Early Intervention Group (Residents) vs Delayed Intervention Group (Residents); We conducted a superiority statistical test to assess if residents' OSCE performance improved after exposure to the PACTS curriculum. OSCE performance was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups. We compared the difference in the percentage of residents designated "mostly" and "a great deal" on Trust and Pain; Test type: Superiority; p = 0.0001, Chi-squared; difference in the percentage = 6.2

6. Secondary Outcome: Patients' Self-reported Satisfaction Scores
Description: We used an adapted version of the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS) to assess patients' (1) satisfaction with pain management, (2) satisfaction with communication including specific measures for limited English proficiency (LEP), (3) trust, and (4) comprehension of informed consent. Patient satisfaction was captured using a modified Likert scale from lowest to highest: strongly disagree, disagree, neither agree nor disagree, agree, and strongly agree. The values reported below are the percentage of participants who reported "agree" or "strongly agree."
Time Frame: Period 2 (18 months)
Population: Patient reported satisfaction surveys at Periods 2 (18 months). Of the 1297 patients in the Early Intervention Group, and 1198 patients in the Delayed Intervention Group, only 436 patients and 392 patients, respectively, completed the survey at Period 2.
Measure: Number; unit: percentage of participants
Groups:
- Early Intervention Group: The investigators will evaluate patient reported satisfaction amongst patients who were cared for my residents who received the PACTS curriculum. Evaluation will be performed at time Period 2 (18 months). Patients designated to the Early Intervention Group were cared for by a resident enrolled in the Early Intervention Group.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group: The investigators will evaluate patient reported satisfaction amongst patients who were cared for by residents who had received the standard residency curriculum. Patients designated to the Delayed Intervention Group were cared for by a resident enrolled in the Delayed Intervention group.
Arm/Group | Early Intervention Group | Delayed Intervention Group
Number analyzed (Participants) | 436 | 392
percentage of participants
  Trust Period 2 | 72.06 | 75.25
  Limited English Proficiency Period 2 | 53.48 | 51.56
  Consent Period 2 | 77.94 | 82.7
  Pain Period 2 | 81.0 | 81.19
Statistical Analysis 1: Comparison: Early Intervention Group vs Delayed Intervention Group; We conducted a superiority statistical test to assess if patient satisfaction improved after resident exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum, patient satisfaction was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups. We compared the difference in proportion of patients who reported "agree" and "strongly agree" for satisfaction as it relates to trust at time period 2; Test type: Superiority; p = 0.5079, Chi-squared; absolute difference between percentage = 3.19
Statistical Analysis 2: Comparison: Early Intervention Group vs Delayed Intervention Group; We conducted a superiority statistical test to assess if patient satisfaction improved after resident exposure to the PACTS curriculum. For purposes of measuring an effect of the curriculum, patient satisfaction was compared at Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups. We compared the difference in proportion of patients who reported "agree" and "strongly agree" for satisfaction as it relates to limited English proficiency at period 2; Test type: Superiority; p = 0.1571, Chi-squared; absolute difference between percentage = 1.92
Statistical Analysis 3: Comparison: Early Intervention Group vs Delayed Intervention Group; We conducted a superiority statistical test to assess if patient satisfaction improved after resident exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum, patient satisfaction was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups. We compared the difference in proportion of patients who reported "agree" and "strongly agree" for satisfaction as it relates to consent at time period 2; Test type: Superiority; p = 0.0001, Chi-squared; absolute difference between percentage = 4.76
Statistical Analysis 4: Comparison: Early Intervention Group vs Delayed Intervention Group; We conducted a superiority statistical test to assess if patient satisfaction improved after resident exposure to the PACTS curriculum. For purposes of measuring an effect of the PACTS curriculum, patient satisfaction was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups. We compared the difference in proportion of patients who reported "agree" and "strongly agree" for satisfaction as it relates to pain at time period 2; Test type: Superiority; p = 0.2956, Chi-squared; absolute difference between percentage = 0.19

7. Secondary Outcome: Median Hospital Length of Stay for Patient Participants
Description: National Surgical Quality Improvement Program (NSQIP) metrics for each patient participant capturing hospital length of stay in days. Patients designated to Early Intervention Group were cared for by a resident enrolled in the Early Intervention group, where the PACTS curriculum was administered between period 1 (0 months) and period 2 (18 months). Patients designated to the Delayed Intervention group were cared for by a resident enrolled in the Delayed Intervention group, where the standard curriculum was administered between period 1 (0 months) and period 2 (18 months). We are comparing median length of stay at period 2.
Time Frame: Period 2 (18 months)
Population: Comparison of length of stay for patients admitted to the hospital and cared for by residents in the early versus delayed intervention groups. The analysis population differs from the overall number of patients because not all patients had a recorded length of stay. Of those that we had length of stay data for, there were 255 participants in the Early Intervention group at Period 2, and 386 participants in the Delayed Intervention group at Period 2.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Early Intervention Group (Patients): The investigators will conduct after the PACTS curriculum at time Period 2 (18 months).
  These data are from patients who are cared for by residents enrolled in the Early Intervention Group at time Period 2.
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group (Patients): The investigators will conduct testing after the standard residency curriculum at time Period 2 (18 months). These data are from patients who are cared for by residents enrolled in the Delayed Intervention Group.
Arm/Group | Early Intervention Group (Patients) | Delayed Intervention Group (Patients)
Number analyzed (Participants) | 255 | 386
Days | 8.85 [5.35 to 12.35] | 14.16 [8.66 to 19.66]
Statistical Analysis 1: Comparison: Early Intervention Group (Patients) vs Delayed Intervention Group (Patients); We conducted a superiority statistical test to assess if patients length of stay improved after resident exposure to the PACTS curriculum. Patient length of stay was compared at time Period 2 between the Early Intervention ("intervention") and Delayed Intervention ("control") groups to measure an effect of the PACTS intervention; Test type: Superiority; p = 0.0028, Wilcoxon (Mann-Whitney); Cox Proportional Hazard = 5.31 — We used Cox Proportional Hazard to assess time to discharge, with 5.31 days as the estimated value for the difference between the two groups

ADVERSE EVENTS:
Time Frame: The entirety of the trial was 36 months, divided into 3 periods: period 1 (0 months), period 2 (18 months), and period 3 (36 months).
Description: Our definition of an adverse event is consistent with that of clinical trials.gov. Our trial did not involve more than a minimal-risk intervention.
Groups:
- Early Intervention / Retention Group, Residents: Residents in the Early Intervention Group undergo baseline assessment at period 1 (0 months) followed by the PACTS curriculum, with subsequent assessment at period 2 (18 months) and period 3 (36 months).
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Delayed Intervention Group, Residents: Residents in the Delayed Intervention Group undergo baseline assessment at period 1 (0 months) followed by the standard curriculum, with subsequent assessment at period 2 (18 months). They then receive the PACTS curriculum with subsequent evaluation at period 3 (36 months).
  PACTS curriculum: The cultural dexterity curriculum, known as PACTS (Provider Awareness Cultural Dexterity Toolkit for Surgeons) focuses on developing cognitive skills to adapt to individual patients' needs to ensure personal, patient-centered surgical care.
  The curriculum is comprised of four educational modules on establishing trust in the physician-patient relationship, communicating effectively with patients with limited English proficiency, discussing informed consent, and issues surrounding pain management. Each module consists of an independent learning activity, an interactive role-play, and a post-lesson assessment.
- Early Intervention Group, Patients: This corresponds to patients who were cared for by residents who were designated to the Early Intervention Group.
- Delayed Intervention Group, Patients: This corresponds to patients who were cared for by residents who were designated to the Delayed Intervention Group.
Arm/Group | Early Intervention / Retention Group, Residents | Delayed Intervention Group, Residents | Early Intervention Group, Patients | Delayed Intervention Group, Patients
All-Cause Mortality (participants affected / at risk) | 0/192 | 0/214 | 0/1297 | 0/1198
Serious Adverse Events (participants affected / at risk) | 0/192 | 0/214 | 0/1297 | 0/1198
Other Adverse Events (participants affected / at risk) | 0/192 | 0/214 | 0/1297 | 0/1198

LIMITATIONS AND CAVEATS:
Duration of trial was impacted by the COVID-19 pandemic, leading to prolonged enrollment time (36 months) as opposed to intended 18 month study duration. Educational interventions and assessments were modified to a virtual platform.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-09-18): https://cdn.clinicaltrials.gov/large-docs/95/NCT03576495/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT03576495/SAP_001.pdf
  • Informed Consent Form (2023-03-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT03576495/ICF_002.pdf